CLINICAL TRIAL: NCT07376941
Title: The Effect of Virtual Reality Distraction on Pain and Discomfort Associated With Bitewing Radiographs in Pediatric Patients
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdulaziz University (Other)
Responsible Party: Principal Investigator, Sara Mustafa Bagher, Associate Professor, King Abdulaziz University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: KingAbdulazizU
Record Dates: First submitted 2026-01-05; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Objective Pain and Discomfort; Subjective Pain and Discomfort; Behavior; Satisfaction; Future Preferences
Keywords: Satisfaction, Virtual Reality, Bitewings Radiographs
MeSH Terms: conditions — Behavior; Personal Satisfaction

STUDY DESIGN:
Intervention Model Description: In the test group, subjects wore VR goggles (LG 360G Electronics) connected to a mobile phone, and a VR headset; the selected video was played. In the control group, BWS were taken without the use of any distraction device.
Who Masked: Outcomes Assessor
Masking Description: Due to the nature of the study, neither the subject nor the radiologist will be blinded to the group allocation. However, the statistician will be blinded to which group each subject will be allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- In the test group, the subjects will wear VR device goggles. (Experimental): In the test group, the subjects will wear VR device goggles (LG 360 virtual reality [VR] headset, LG Electronics) connected to a mobile phone, and the chosen video will be played.
  Interventions: Other: virtual reality device goggles
- In the control group, radiographs will be taken without the use of any distraction device. (No Intervention): In the control group, radiographs will be taken without the use of any distraction device.

INTERVENTIONS:
Other: virtual reality device goggles — virtual reality device goggles (LG 360 virtual reality [VR] headset, LG Electronics)
  Arms: In the test group, the subjects will wear VR device goggles.

SUMMARY:
This study will be conducted at King Abdulaziz University Dental Hospital (KAUDH). Ethical approval was obtained from the Research Ethics Committee of the Faculty of Dentistry at King Abdulaziz University (32-03-25).

Inclusion criteria will include healthy and cooperative children aged 4 to 12 years who are referred to the radiology department for two-bitewing radiographs. Children with a history of epilepsy or anxiety disorder will be excluded. The study's purpose, risks, benefits, and limitations will be explained to the parents or guardians of eligible children by trained dental interns. Those who agree to participate will be asked to sign an Arabic consent form before their involvement. Additionally, an assent form will be obtained from children aged seven and older.

Subjects' age, gender, previous dental experience, and behavior during previous dental visits, as assessed by Frankl's behavior rating scale , will be recorded, along with whether they own or have prior exposure to a virtual reality device. Only children with cooperative and definitely cooperative behavior will be included.

A randomization sequence with an allocation ratio of 1:1 will be generated using computer software and kept with a radiology assistant who is not involved in the study to ensure allocation concealment. Due to the nature of the study, neither the subject nor the radiologist will be blinded to the group allocation. However, the statistician will be blinded to which group each subject will be allocated.

Before taking the radiographs, subjects will be asked to select a video from a list of popular cartoon shows or a video of their preference. In the test group, the subjects will wear virtual reality device goggles (LG 360 virtual reality [VR] headset, LG Electronics) connected to a mobile phone, and the chosen video will be played. In the control group, radiographs will be taken without the use of any distraction device. The sounds of the videos will be played on headphones. All bitewing radiographs will be taken by the same radiologist, following the As Low As Reasonably Achievable (ALARA) protocol and hospital guidelines. The procedure uses either size one or size two bitewing Photostimulable Phosphor digital sensors, along with a film holder and a rectangular collimator. While taking the radiographs, the Tell-Show-Do behavior management technique will be used with all participating children, and they will be recorded with a high-resolution camera.

The camera will aim toward the face and the body. Later, two trained and calibrated evaluators will independently assess the participating children's behavioral pain using the face, legs, activity, cry, and consolability (FLACC) behavioral pain assessment scale. The FLACC scale ranges from 0 to 10, with 0 indicating no pain and 10 the worst possible pain. Additionally, the behavior during the BWS will also be recorded using Frankl's behavior rating scale classification. Training and calibration for the evaluators will involve watching videos of 20 randomly selected children during their dental treatment. A stopwatch will be used to measure the chair time required to take the radiographs. In the test group, the time needed to place the VR device will be included.

Immediately after taking the BWS, the subjects will be shown the Arabic version of the Wong-Baker FACES pain rating scale. They will be asked to select the face that best describes their feelings during the procedure. Finally, the satisfaction with the use of VR during BWS taking will be assessed using a five-point Likert scale, where zero indicates 'not satisfied at all' and 10 means' very satisfied'. Subjects who require repeating any of the BWS will be excluded from the study

ELIGIBILITY:
Inclusion Criteria:

1. Healthy
2. Cooperative children
3. Aged 4 to 12 years
4. Referred to the radiology department for two-bitewing radiographs.

Exclusion Criteria:

1- Children with a history of epilepsy or anxiety disorder

Ages: 4 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-05-30 (Estimated); Study Completion 2026-05-30 (Estimated)

PRIMARY OUTCOMES:
Objective main and discomfort | While taking the BWS radiographs.
  The camera will aim toward the face and the body. Later, two trained and calibrated evaluators will independently assess the participating children's behavioral pain using the FLACC scale. The FLACC scale ranges from 0 to 10, with 0 indicating no pain and 10 the worst possible pain.
Subjective pain and discomfort | Immediately after taking the BWS.
  Immediately after taking the BWS, the subjects will be shown the Arabic version of the Wong-Baker FACES pain rating scale. They will be asked to select the face that best describes their feelings during the procedure. The participants choose the face that best describes their current feelings, ranging from 0 (no hurt) to 10 (worst pain).

SECONDARY OUTCOMES:
The behavior during the radiograph procedure. | While taking the BWS radiographs
  The camera will aim toward the face and the body. Later, two trained and calibrated evaluators will independently assess the participating children's behavior during the radiograph procedure will also be recorded using Frankl's behavior rating scale classification
Satisfaction of the use of virtual reality | Immediately after taking the BWS
  The satisfaction with the use of VR during radiograph taking will be assessed using a five-point Likert scale, where zero indicates 'not satisfied at all' and 10 means' very satisfied'.

CONTACTS AND LOCATIONS:
Locations (1):
- King Abdulaziz Univeristy, Jeddah, Saudi Arabia

IPD SHARING:
Plan to Share IPD: No